CLINICAL TRIAL: NCT01741948
Title: Hormonal Contraceptive Use and the Risk of Provoked Vestibulodynia- A Prospective Study
Brief Title: Hormonal Contraceptive Use and the Risk of Provoked Vestibulodynia
Status: Withdrawn | Type: Observational
Why Stopped: the study has never started. my grant request was denied.
Sponsor: ahinoam lev sagie (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor-Investigator, ahinoam lev sagie, Principal Investigator, Clalit Health Services
Organization: Clalit Health Services (Other)
Other Study IDs: Levsagie OCP PVD
Record Dates: First submitted 2012-11-23; First posted 2012-12-05 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Vestibulodynia
Keywords: Provoked vestibulodynia; Hormonal contraceptives
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood cells will be extracted from all blood samples. mRNA will be purified from all samples. The mRNA will be divided to aliquots and will be frozen in -80°C until further processing after all cohort samples have been collected.
  mRNAs will be purified from whole blood using the QIAamp RNA purification kit (Quiagen Germany). A DNase I (Qiagen) digestion step is included in order to eliminate genomic DNA.
  Serum will be collected from all blood samples. It will will be frozen in -70°C until further processing after all cohort samples have been collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First time users of hormonal contraceptive
  Interventions: Drug: Hormonal contraceptive

INTERVENTIONS:
Drug: Hormonal contraceptive — The study will follow patients who are first time users of HCs for a full year after initiation. Patients will be followed every 3 months via questionnaires, blood examinations, and gynecologic examination, in case dyspareunia evolves.
  First appointment (before initiation of HCs):
  Questionnaire FSFI (Female Sexual Function Index) questionnaire. Blood collection for hormones levels and extraction of mononuclear blood cells. A gynecologic exam intended to rule out existing problem which causing dyspareunia.
  3,6,9,and 12 months after initiation of HCs or anytime if a patient has dyspareunia:
  Questionnaire evaluating possible influence of HCs use (dyspareunia, lubrication and libido).
  FSFI questionnaire. Blood collection Gynecologic examination, designated to assess the cause of pain, including assessment of vestibular tenderness, muscle tightness and tenderness, pressure-pain thresholds measurement using vulvar algesiometer, pH measurement and vaginal swab for microscopy.

SUMMARY:
There have been reports in the medical literature demonstrating a link between the development of provoked vestibulodynia (PVD), a sexual pain disorder, and hormonal contraceptive (HC) use. The purpose of this pilot study is to assess the prevalence of HCs induced PVD among a HC naïve population, to evaluate which of the components of the HCs are associated with a higher risk of the development of PVD, and to evaluate which clinical and genetic factors predispose the patient to HCs induced PVD. Assessments will be made through patient questionnaires, physical examinations, and blood tests. Microarray techniques will be employed to characterize, on a global level, the gene expression profiles of women who develop PVD in comparison to those who do not develop PVD. Patients will be followed for a year. Results will be used to develop a larger clinical trial.

DETAILED DESCRIPTION:
Background:

Provoked vestibulodynia (PVD), previously called vulvar vestibulitis syndrome, is clinically defined as chronic, unexplained, vulvar pain or discomfort, confined to the vulvar vestibule, in response to contact or pressure. As a result, women with PVD experience pain on sexual intercourse, and many patients also have pain in response to non-sexual activities. The actual prevalence of PVD is unknown, but current evidence indicates that the lifetime cumulative incidence of vulvodynia approaches 15%. Currently, PVD is thought to be the leading cause of dyspareunia in premenopausal women. Once a woman with PVD develops the syndrome, symptoms may last for years; as a result, PVD has a profound effect on women's sexuality and psychological well-being.

The diagnosis of PVD is usually made by assessing for the presence of the modified Friedrich's criteria. These criteria consist of 1) a history of vulvar pain, dyspareunia or pain with tampon insertion, 2) tenderness of the vestibule when being touched with a cotton-tip applicator, and 3) no other identifiable cause for the pain (such as vaginitis, dermatitis etc.).

The etiology of this condition remains unknown. Proposed causes include chronic inflammation, peripheral neuropathy, genetic, immunologic and\or hormonal factors, infection, psychological disorders, sexual dysfunction, or disturbance in the central nervous system.

Several studies have demonstrated an increased risk of developing PVD secondary to hormonal contraceptive (HC) usage. The relative risk of developing PVD seems to rise with an increased duration of HCs use (at least up to 2-4 years of use), first use of HCs at a young age (<16 years), and the hormonal composition of HCs, specifically the progestogenic, estrogenic, and androgenic potency of the pills.

Several mechanisms of action have been suggested for HCs induced PVD:

* Alteration of vestibular hormonal receptors.
* Alterations of the morphological pattern of the vestibular mucosa(13).
* Decreased pain threshold.
* Alteration of serum free hormones levels.

Objectives/Purpose of the Study:

1. To assess the actual prevalence of HCs induced PVD in a prospective study.
2. To evaluate which of the components contained in the HCs (oral contraceptives, transdermal patch, vaginal ring) are associated with higher risk of HCs induced PVD, specifically; the dose of ethinyl estradiol (15, 20 and 30 mcg) and the progesterone component.
3. To evaluate which factors predispose the patient to HCs induced PVD. We will analyze both clinical (age, age at menarche, length of use, body mass index etc.), hormonal (E2, testosterone etc.) and altered gene expression factors.

The proposed study is a preliminary investigation aimed at estimating the rate of HCs induced PVD. The data from this study will enable the determination of the number of patients needed to obtain statistical significance in a future, larger study regarding patients' risk factors for developing PVD and HCs formulation.

For this pilot study the investigators will evaluate 200 patients and follow them for a total of 1 year after HC initiation. Since this is a novel study that has not been investigated, nor is there available statistics in the medical literature, the investigators anticipate that 200 patients will provide enough data regarding incidence of PVD development secondary to HCs use.

Definitions and measures to be used to diagnose HC induced PVD:

1. New onset of vulvar pain suggestive of PVD, i.e. symptoms of pain on vaginal penetration (insertional dyspareunia and/or pain with tampon insertion), following initiation of HCs.
2. On exam, tenderness localized within the vestibule when being touched with a cotton-tip applicator. The exam will be performed on defined points of the labia minora, labia majora and the vestibule in 5 defined points (1,5,6,7,11), with patients reporting pain verbally by a rating scale of 0 to 10 at each point.
3. No identifiable cause for the pain, such as vulvovaginal candidiasis, desquamative inflammatory vaginitis (DIV), herpes, dermatitis or vulvar dystrophy.

Time frame for completion: The investigators anticipate one year for patients' enrollment and another year for follow up. Data analysis and microarray analyses will be done during the third year. Data should be available within 3 years of study initiation.

ELIGIBILITY:
Inclusion Criteria:

* 200 non pregnant women between 18-35 naïve to HCs or other hormonal medications.
* Patients able to provide Informed Consent and complete questionnaires.
* Patient intends to use HCs for at least one year.
* On exam before initiation of HCs, patient does not have primary PVD, pelvic floor hypertonicity, vaginismus or congenital abnormalities.
* Patient will be available for follow up appointments.
* Patient is willing to undergo gynecologic examination, if dyspareunia develops.

Exclusion Criteria:

* Patients with endocrine disturbances (including PCOS), liver diseases and eating disorders.
* Patients who suffer from Hypertension, Migraine with aura or clotting disturbances.
* Patients that experience pain with intercourse or tampon insertion.
* Patients that have other contraindications for HCs use

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will follow patients who are first time users of HCs for a full year after initiation. Patients will be recruited in a gynecology clinic affiliated with the "Clalit" Health Maintenance Organization in Jerusalem, Israel (Merkaz Briut Haisha, Ramat Eshkol, Jerusalem). This is a primary care government funded clinic, treating a diverse population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of hormonal-contraceptive induced provoked vestibulodynia | One year
  one year for patients' enrollment and another year for follow up.

SECONDARY OUTCOMES:
Hormonal contraceptive components associated with higher risk of HCs induced PVD | One year
  Dose of ethinyl estradiol (15, 20 and 30 mcg) The progesterone component
Clinical factors associated with HCs induced PVD | One year
  Age at menarche Length of use Body mass index
Biochemical markers associated with higher risk of HCs induced PVD | One year
  Hormones: E2, testosterone Altered gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam LevSagie, MD, Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Clalit health Services, Jerusalem
  - Hadassah Medical Organization, Jerusalem

REFERENCES:
- [Background] Goldstein A, Burrows L, Goldstein I. Can oral contraceptives cause vestibulodynia? J Sex Med. 2010 Apr;7(4 Pt 1):1585-7. doi: 10.1111/j.1743-6109.2009.01685.x. Epub 2010 Jan 25. PMID 20102483
- [Background] Greenstein A, Ben-Aroya Z, Fass O, Militscher I, Roslik Y, Chen J, Abramov L. Vulvar vestibulitis syndrome and estrogen dose of oral contraceptive pills. J Sex Med. 2007 Nov;4(6):1679-83. doi: 10.1111/j.1743-6109.2007.00621.x. PMID 17970976
- [Background] Bohm-Starke N, Johannesson U, Hilliges M, Rylander E, Torebjork E. Decreased mechanical pain threshold in the vestibular mucosa of women using oral contraceptives: a contributing factor in vulvar vestibulitis? J Reprod Med. 2004 Nov;49(11):888-92. PMID 15603099
- [Background] Bouchard C, Brisson J, Fortier M, Morin C, Blanchette C. Use of oral contraceptive pills and vulvar vestibulitis: a case-control study. Am J Epidemiol. 2002 Aug 1;156(3):254-61. doi: 10.1093/aje/kwf037. PMID 12142260
- [Background] Sjoberg I, Nylander Lundqvist EN. Vulvar vestibulitis in the north of Sweden. An epidemiologic case-control study. J Reprod Med. 1997 Mar;42(3):166-8. PMID 9109085
- [Background] Bazin S, Bouchard C, Brisson J, Morin C, Meisels A, Fortier M. Vulvar vestibulitis syndrome: an exploratory case-control study. Obstet Gynecol. 1994 Jan;83(1):47-50. PMID 8272306
- [Background] Johannesson U, Sahlin L, Masironi B, Hilliges M, Blomgren B, Rylander E, Bohm-Starke N. Steroid receptor expression and morphology in provoked vestibulodynia. Am J Obstet Gynecol. 2008 Mar;198(3):311.e1-6. doi: 10.1016/j.ajog.2007.09.041. Epub 2008 Feb 21. PMID 18177837
- [Background] Johannesson U, Sahlin L, Masironi B, Rylander E, Bohm-Starke N. Steroid receptor expression in the vulvar vestibular mucosa--effects of oral contraceptives and menstrual cycle. Contraception. 2007 Oct;76(4):319-25. doi: 10.1016/j.contraception.2007.06.014. Epub 2007 Aug 28. PMID 17900445
- [Background] Johannesson U, Blomgren B, Hilliges M, Rylander E, Bohm-Starke N. The vulval vestibular mucosa-morphological effects of oral contraceptives and menstrual cycle. Br J Dermatol. 2007 Sep;157(3):487-93. doi: 10.1111/j.1365-2133.2007.08066.x. Epub 2007 Jul 11. PMID 17627793
- [Background] Eva LJ, MacLean AB, Reid WM, Rolfe KJ, Perrett CW. Estrogen receptor expression in vulvar vestibulitis syndrome. Am J Obstet Gynecol. 2003 Aug;189(2):458-61. doi: 10.1067/s0002-9378(03)00365-x. PMID 14520218
- [Background] Harlow BL, Vitonis AF, Stewart EG. Influence of oral contraceptive use on the risk of adult-onset vulvodynia. J Reprod Med. 2008 Feb;53(2):102-10. PMID 18357801
- [Background] Harlow BL, Stewart EG. A population-based assessment of chronic unexplained vulvar pain: have we underestimated the prevalence of vulvodynia? J Am Med Womens Assoc (1972). 2003 Spring;58(2):82-8. PMID 12744420